CLINICAL TRIAL: NCT01318421
Title: An Open-Label, Long-Term, Follow-Up Study of Subcutaneous ELND002 in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: A Study of ELND002 in Patients With Relapsing Forms of Multiple Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELND002-MS153
Record Dates: First submitted 2011-03-08; First posted 2011-03-18 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing forms of secondary progressive multiple sclerosis (SPMS)or relapsing-remitting multiple sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ELND002 (Experimental): ELND002 sc injection
  Interventions: Drug: ELND002

INTERVENTIONS:
Drug: ELND002

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of ELND002 in patients with multiple sclerosis (MS) after participation in study MS103.

ELIGIBILITY:
Inclusion Criteria:

* This study is open only to subjects who have completed the week 12 visit in study ELND002-MS103 while taking their assigned dose of study drug.

Exclusion Criteria:

* Subject has no new medical contraindications to continue participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of ELND002 including the identification of dose-limiting toxicity(ies) (DLT). | 1 year
  Safety and tolerability will be assessed by frequency and severity of AEs.

SECONDARY OUTCOMES:
To evaluate the PK/PD/BM measurement of ELND002 in patients with MS. | 1 year
  Measurement of drug concentration, alpha 4 receptor saturation, soluble VCAM and MADCAM.